CLINICAL TRIAL: NCT04847596
Title: An Open-label Multicenter Single-arm Pilot Study to Assess Immune Response to COVID-19 Vaccine in Participants With Relapsing Multiple Sclerosis Treated With Ofatumumab 20 mg Subcutaneously
Brief Title: A Multicenter Study to Assess Response to COVID-19 Vaccine in Multiple Sclerosis Participants Treated With Ofatumumab
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GUS18
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: COVID-19; vaccine; ofatumumab; SARS-coV2; antibody; open-label
MeSH Terms: conditions — COVID-19 | interventions — ofatumumab; COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- participants with RMS treated with ofatumumab: Relapsing MS participants receiving a full course (two doses) of a COVID-19 mRNA vaccine after starting ofatumumab 20 mg subcutaneous treatment
  Interventions: Other: Ofatumumab; Other: Covid-19 vaccine

INTERVENTIONS:
Other: Ofatumumab — Prospective observational cohort study. There is no treatment allocation. Patients administered Ofatumumab by prescription that have started before inclusion of the patient into the study will be enrolled.
Other: Covid-19 vaccine — Prospective observational cohort study. There is no treatment allocation. Participants will obtain the COVID-19 FDA approved Emergency Use mRNA vaccine through their HCP (private insurance) or appropriate federal, state or local program.

SUMMARY:
This is a single arm, pilot multicenter prospective study in up to 22 participants with relapsing multiple sclerosis. Patients screened for the study can either be scheduled for vaccine, have received a single vaccine with a scheduled second dose, or already completed full course (two dose) vaccination. Fully vaccinated participants must be able to complete immune assay No.1 ≥ 14 days after the second dose of vaccine

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Age 18-55 years old inclusive at Screening
3. Diagnosis of relapsing MS by 2017 revised McDonald criteria
4. Must be willing to comply with the study schedule
5. Have received/scheduled vaccination with a FDA approved for emergency use COVID-19 mRNA vaccine (either Pfizer or Moderna) (i) either been scheduled for vaccine, (ii) received a single vaccine with a scheduled second dose, or (iii) already completed full course (two dose) vaccination.
6. Currently receiving ofatumumab for the treatment of RMS (Preoftumumab serology with Hepatitis B testing showing no active or latent infection, as well as serum IgG results to be recorded in the database if available)

Exclusion Criteria:

1. Known clinical diagnosis of COVID-19 prior to screening based on investigator's or patient's personal physician's judgement
2. Has a contraindication to receiving an mRNA COVID-19 vaccine
3. Has an immediate allergic reaction to past vaccine or injection
4. Any safety finding including low IgG and/or low IgM levels requiring an ofatumumab treatment interruption within the 12 weeks immediately prior to vaccination as determined by the HCP
5. Any major episode of infection requiring hospitalization or treatment with intravenous antibiotics within 2 weeks prior to the screening visit
6. Prior treatment with S1P agent within 2 months of study enrollment
7. Prior treatment with natalizumab within 6 months of study enrollment
8. Contraindications to ofatumumab treatment as per the USPI will be adhered to which include active infection hepatitis B infection, progressive multifocal leukoencephalopathy and pregnancy.
9. Participation in another interventional clinical trial within 14 days before enrollment.
10. Have been treated with any of the medications as described in the full protocol
11. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for 6 months after stopping medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Relapsing MS participants receiving a full course (two doses) of a COVID-19 mRNA vaccine after starting ofatumumab 20 mg subcutaneous treatment
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving immune response - immune assay No. 1 | 14 days after full course vaccination (two doses)
  Achieving immune response as defined by a positive SARS-CoV-2 qualitative IgG antibody assay. (yes/no)

SECONDARY OUTCOMES:
Proportion of participants achieving immune response - immune assay No. 2 | 90 days post assay 1
  Achieving immune response as defined by a positive SARS-CoV-2 qualitative IgG antibody assay 90 days after assay No. 1 (yes/no)
Adverse events/serious adverse events | 120 days after full course vaccination
  An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
  Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (4):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Owosso, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Plainview, New York
- Novartis Investigative Site, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bar-Or A, Aburashed R, Chinea AR, Hendin BA, Lucassen E, Meng X, Stankiewicz J, Tullman MJ, Cross AH. Humoral immune response to COVID-19 mRNA vaccines in patients with relapsing multiple sclerosis treated with ofatumumab. Mult Scler Relat Disord. 2023 Nov;79:104967. doi: 10.1016/j.msard.2023.104967. Epub 2023 Aug 28. PMID 37769429
- See also: Results for COMB157GUS18 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18009